CLINICAL TRIAL: NCT07211620
Title: KInetics of Procalcitonin to Reduce Unnecessary aNtibiotic Use (KIPRUN) - Protocol for a Multi-center, Randomized, Superiority Trial to Compare the Efficacy and Safety of Procalcitonin Kinetics-guided and Absolute Procalcitonin Value-guided Antibiotic Initiation in Reducing Unnecessary Antibiotic Therapy in Critically Ill Patients
Brief Title: KInetics of Procalcitonin to Reduce Unnecessary aNtibiotic Use - Comparing Procalcitonin Kinetics-guided and Absolute Procalcitonin Value-guided Antibiotic Initiation in Reducing Unnecessary Antibiotic Use in Critically Ill Patients
Acronym: KIPRUN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Dr. Papp Márton, co-head of the unit, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: BM/20019- 1/2025
Record Dates: First submitted 2025-09-21; First posted 2025-10-08 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-09

CONDITIONS: Infection; Sepsis
Keywords: procalcitonin; bacterial infection; antibiotics; kinetics
MeSH Terms: conditions — Infections; Sepsis; Bacterial Infections | interventions — Kinetics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Nurses
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinetics (Experimental): In the case of a suspected new-onset infection, the treating physician starts antibiotic therapy according to a predefined protocol depending on the kinetics of PCT.
  Interventions: Other: Kinetics
- Absolute (Experimental): In the case of a new-onset infection, starting ABs is recommended depending on the actual absolute value of PCT.
  Interventions: Other: Absolute

INTERVENTIONS:
Other: Kinetics — Initiation of the AB therapy is recommended for the clinician if PCT ≥ 0.5 ng/ml and PCT elevation ≥100% from the previous day's value.
  Arms: Kinetics
Other: Absolute — According to the antibiotic protocol, starting ABs is recommended if PCT ≥ 0.5 ng/ml.
  Arms: Absolute

SUMMARY:
The study aims to compare the efficacy and safety of an absolute procalcitonin (PCT) value-guided antibiotic initiation protocol and a protocol using the kinetics of PCT (the difference between the actual and the previous day value) in hemodynamically stable critically ill patients with suspected new-onset infection on admission or during ICU stay.

The main question it aims to answer:

* Can the investigators decrease the number of unnecessary AB therapies using the kinetics of PCT insted of using absolute PCT values?
* Is it safe to use PCT kinetics together with the clinical picture to guide AB initiation? AB therapy will be initiated according to predefined PCT protocols (Kinetics and Absolute Group). After 72 hours of treatment, an independent multidisciplinary team (infectologist, microbiologist and intensivist) will decide about the necessity of the treatment with all the relevant results in hand.

DETAILED DESCRIPTION:
Appropriate antibiotic (AB) therapy is still a big challenge in intensive care units today. More than 50% of our patients are considered potentially infected, and infection alone can double mortality; however, infection is later confirmed in less than 60% of patients admitted with the initial diagnosis of sepsis. According to previous studies, at least every fifth patient in intensive care units receives unnecessary antibiotics (ABs), leading to the well-known adverse effects of ABs without any benefit. The emergence of AB resistance has been associated with 700,000 avoidable deaths in 2014, and WHO estimates that it will contribute to the death of 10 million people by 2050.

Procalcitonin (PCT) is one of the most studied inflammatory biomarkers. Several randomized controlled trials (RCTs) and their meta-analyses concluded that PCT-guided antibiotic treatment could reduce the length of AB therapy without adverse effects; moreover, it may be associated with reduced 28-day mortality, which was also confirmed by our study in 2023. Accordingly, the current sepsis guideline recommends the combined evaluation of the clinical picture and PCT when stopping AB therapy; however, it contains a weak recommendation against using PCT when starting the treatment. The latter proposition is based on three studies with a significant number of surgical patients (around 40%) in two of them, in whom the applied PCT cut-off (0.5-1 ng/ml) presumably was too low, supported by several previous studies. Therefore, the overuse of ABs was more or less hardcoded into the protocol.

Kinetics of an inflammatory biomarker can carry much more information about the host response to infection instead of a single value. In a prospective observational study by Trasy et al., early PCT kinetics (PCT change between the day of suspected infection and the previous 24 hours) predicted infection, while PCT did not change in the group of patients in whom the infection was later ruled out. Tsangaris and his colleagues measured PCT daily in critically ill patients. The investigators noted a two-fold increase in PCT levels between the day of fever onset and the previous day if the patients had an infection, while there was no difference in the PCT values if the participants had no infection.

Based on these findings, the investigators created a protocol to reduce the number of unnecessary antibiotic therapies using the kinetics of PCT.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years < ) non-surgical, surgical, or trauma patients
* Suspected new-onset infection on admission or during ICU stay
* The source of infection is known or highly suspected, and source control has been implemented if needed (i.e., removal of an infected device (e.g., central line, endoprosthesis)
* Two PCT values are available - one on the day of suspicion of infection and one 24±4 hours earlier.
* Microbiology sampling has to be performed (according to all presumed sources - blood culture -aerobic and anaerobic, lower respiratory tract sample (tracheal aspirate/bronchoalveolar lavage), urine, etc.).
* Written informed consent of the patient (or legal guardian if the patient cannot provide consent)

Exclusion Criteria:

* Septic shock (hypotension requiring vasopressor therapy to maintain mean blood pressure of 65 mmHg or greater and having a serum lactate level greater than 2 mmol/L after adequate fluid resuscitation)
* Infections for which long-term antibiotic treatment is strongly recommended (e.g., infective endocarditis, osteoarticular infections, chronic prostatitis, tuberculosis)
* Infections related to primary surgical intervention and adequate source control cannot be guaranteed (e.g., fecal peritonitis, pancreatic necrosectomy, infective necrotizing fascitis - i.e., Fournier's gangrene),
* Indisputable infections (e.g., hepatic abscess, empyema)
* Poor chance of survival (i.e., expected ICU stay less than 24 hours or initial Acute Physiology and Health Evaluation Score II (APACHE II) >30)
* Admissions after cardiopulmonary resuscitation
* Severe immunosuppression other than steroid use
* stem-cell transplant recipients
* solid organ transplant patients
* HIV infection with a CD4 count of less than 200 cells/mm3
* Neutropenia with less than 500 neutrophils/mm3
* Patients on ABs within 72 hours before inclusion
* Patients in pregnancy or breastfeeding. Women of childbearing age will be screened by a urine pregnancy test before inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of unnecessary antibiotic therapy | From date of enrollment until 72 hours.
  The number of unjustified antibiotic therapies divided by the number of all therapies.

SECONDARY OUTCOMES:
Organ-support free days | From date of enrollment until the date of disharge of the patient from the ICU or the date of patient's death from any cause, whichever came first, assessed up to 6 months.
  Number of days alive without life support - mechanical ventilation, vasoactive therapy and renal replacement therapy.
Lenght of stay at the intensive care unit | From date of enrollment until the date of discharge of patient from the ICU or the date of patient's death from any cause, whichever came first, assessed up to 6 months.
  Number of days the patient stays at ICU
Length of stay in hospital | From date of enrollment until the date of hospital discharge of the patient or the date of patient's death from any cause, whichever came first, assessed up to 6 months.
  Number of days the patient stays in the hospital
Duration of mechanical ventilation | From date of enrollment until date of ICU discharge of the patient or date of patient's death from any cause, whichever came first, asessed up to 6 months.
  Duration of mechanical ventilation in days
Duration of renal replacement therapy | From date of enrollment until date of hospital discharge of the patient or date of patient's death from any cause, whichever came first, assessed up to 6 months.
  Duration of renal replacement therapy in days
Duration of catecholamine circulatory support | From date of enrollment until date of ICU discharge of the patient or date of patient's death from any cause, whichever came first, assessed up to 6 months.
  Duration of catecholamine circulatory support in days
ICU mortality | From date of enrollment until the date of ICU discharge of the patient, assessed up to 6 months.
  The number of patients died during ICU stay devided by the number of patients enrolled.
28-day mortality | From date of enrollment until day 28.
  The number of patients died divided by the number of patients enrolled.
In-hospital mortality | From date of enrollment until hospital discharge of the patient, assessed up to 6 months.
  The number of patients died devided by the number of patients enrolled.
Number of Multidrug-resistant Organism caused infections | From date of enrollment until the date of hospital discharge of the patient or the patient's death from any cause, whichever came first, assessed up to 6 months.
  Number of diagnosed infections caused by bacteria that are resistant to one or more classes of antimicrobial agents.
Number of Clostridioides difficile infections | From date of enrollment until the date of hospital discharge of the patient or the patient's death from any cause, whichever came first, assessed up to 6 months.
  Number of verified Clostridioides difficile infections

CONTACTS AND LOCATIONS:
Overall Officials: Nikolett Kiss, Study Chair — Semmelweis University; László Zubek, Study Chair — Semmelweis University; Caner Turan, Study Chair — Semmelweis University; Dilan M. Karim, Study Chair — Semmelweis University
Locations (2):
- Hungary (2):
  - Saint Margaret's Hospital, Budapest
  - Semmelweis University, Department of Intensive Therapy, Budapest

IPD SHARING:
Plan to Share IPD: Yes
All data obtained through the study may be provided to researchers with an interest in optimizing antibiotic therapy of critically ill patients. Data and samples will be coded if shared with no protected health information included.
  Zsolt Molnár will receive invitations/requests to share individual participant data, and will consider if the request: 1) explicitly serves public benefit, 2) complies with local ethical and data security regulations of the requesting and providing institutions, 3) lays out the existing or planned legal and technical infrastructure for data transfer, 4) provides a publicly available protocol for planned statistical analyses.

REFERENCES:
- [Background] Shankar-Hari M, Phillips GS, Levy ML, Seymour CW, Liu VX, Deutschman CS, Angus DC, Rubenfeld GD, Singer M; Sepsis Definitions Task Force. Developing a New Definition and Assessing New Clinical Criteria for Septic Shock: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):775-87. doi: 10.1001/jama.2016.0289. PMID 26903336
- [Background] Tsangaris I, Plachouras D, Kavatha D, Gourgoulis GM, Tsantes A, Kopterides P, Tsaknis G, Dimopoulou I, Orfanos S, Giamarellos-Bourboulis E, Giamarellou H, Armaganidis A. Diagnostic and prognostic value of procalcitonin among febrile critically ill patients with prolonged ICU stay. BMC Infect Dis. 2009 Dec 22;9:213. doi: 10.1186/1471-2334-9-213. PMID 20028533
- [Background] Trasy D, Tanczos K, Nemeth M, Hankovszky P, Lovas A, Mikor A, Hajdu E, Osztroluczki A, Fazakas J, Molnar Z. Delta Procalcitonin Is a Better Indicator of Infection Than Absolute Procalcitonin Values in Critically Ill Patients: A Prospective Observational Study. J Immunol Res. 2016;2016:3530752. doi: 10.1155/2016/3530752. Epub 2016 Aug 15. PMID 27597981
- [Background] Szakmany T, Molnar Z. Procalcitonin levels do not predict mortality following major abdominal surgery. Can J Anaesth. 2003 Dec;50(10):1082-3. doi: 10.1007/BF03018387. No abstract available. PMID 14656802
- [Background] Trasy D, Tanczos K, Nemeth M, Hankovszky P, Lovas A, Mikor A, Laszlo I, Hajdu E, Osztroluczki A, Fazakas J, Molnar Z; EProK study group. Early procalcitonin kinetics and appropriateness of empirical antimicrobial therapy in critically ill patients: A prospective observational study. J Crit Care. 2016 Aug;34:50-5. doi: 10.1016/j.jcrc.2016.04.007. Epub 2016 Apr 13. PMID 27288610
- [Background] Najafi A, Khodadadian A, Sanatkar M, Shariat Moharari R, Etezadi F, Ahmadi A, Imani F, Khajavi MR. The Comparison of Procalcitonin Guidance Administer Antibiotics with Empiric Antibiotic Therapy in Critically Ill Patients Admitted in Intensive Care Unit. Acta Med Iran. 2015;53(9):562-7. PMID 26553084
- [Background] Layios N, Lambermont B, Canivet JL, Morimont P, Preiser JC, Garweg C, Ledoux D, Frippiat F, Piret S, Giot JB, Wiesen P, Meuris C, Massion P, Leonard P, Nys M, Lancellotti P, Chapelle JP, Damas P. Procalcitonin usefulness for the initiation of antibiotic treatment in intensive care unit patients. Crit Care Med. 2012 Aug;40(8):2304-9. doi: 10.1097/CCM.0b013e318251517a. PMID 22809906
- [Background] Jensen JU, Hein L, Lundgren B, Bestle MH, Mohr TT, Andersen MH, Thornberg KJ, Loken J, Steensen M, Fox Z, Tousi H, Soe-Jensen P, Lauritsen AO, Strange D, Petersen PL, Reiter N, Hestad S, Thormar K, Fjeldborg P, Larsen KM, Drenck NE, Ostergaard C, Kjaer J, Grarup J, Lundgren JD; Procalcitonin And Survival Study (PASS) Group. Procalcitonin-guided interventions against infections to increase early appropriate antibiotics and improve survival in the intensive care unit: a randomized trial. Crit Care Med. 2011 Sep;39(9):2048-58. doi: 10.1097/CCM.0b013e31821e8791. PMID 21572328
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Hylander Moller M, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock 2021. Crit Care Med. 2021 Nov 1;49(11):e1063-e1143. doi: 10.1097/CCM.0000000000005337. No abstract available. PMID 34605781
- [Background] Papp M, Kiss N, Baka M, Trasy D, Zubek L, Fehervari P, Harnos A, Turan C, Hegyi P, Molnar Z. Procalcitonin-guided antibiotic therapy may shorten length of treatment and may improve survival-a systematic review and meta-analysis. Crit Care. 2023 Oct 13;27(1):394. doi: 10.1186/s13054-023-04677-2. PMID 37833778
- [Background] de Kraker ME, Stewardson AJ, Harbarth S. Will 10 Million People Die a Year due to Antimicrobial Resistance by 2050? PLoS Med. 2016 Nov 29;13(11):e1002184. doi: 10.1371/journal.pmed.1002184. eCollection 2016 Nov. PMID 27898664
- [Background] Montravers P, Dupont H, Gauzit R, Veber B, Bedos JP, Lepape A; Club d'Infectiologie en Anesthesie-Reanimation Study Group. Strategies of initiation and streamlining of antibiotic therapy in 41 French intensive care units. Crit Care. 2011;15(1):R17. doi: 10.1186/cc9961. Epub 2011 Jan 13. PMID 21232098
- [Background] Klein Klouwenberg PM, Cremer OL, van Vught LA, Ong DS, Frencken JF, Schultz MJ, Bonten MJ, van der Poll T. Likelihood of infection in patients with presumed sepsis at the time of intensive care unit admission: a cohort study. Crit Care. 2015 Sep 7;19(1):319. doi: 10.1186/s13054-015-1035-1. PMID 26346055
- [Background] Vincent JL, Sakr Y, Singer M, Martin-Loeches I, Machado FR, Marshall JC, Finfer S, Pelosi P, Brazzi L, Aditianingsih D, Timsit JF, Du B, Wittebole X, Maca J, Kannan S, Gorordo-Delsol LA, De Waele JJ, Mehta Y, Bonten MJM, Khanna AK, Kollef M, Human M, Angus DC; EPIC III Investigators. Prevalence and Outcomes of Infection Among Patients in Intensive Care Units in 2017. JAMA. 2020 Apr 21;323(15):1478-1487. doi: 10.1001/jama.2020.2717. PMID 32207816